CLINICAL TRIAL: NCT06380023
Title: An Investigation Into the Dispersion Pattern During Coughing and Open Nasopharyngeal Suction Using Various Barrier Devices
Status: Completed | Type: Observational
Sponsor: North District Hospital (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TO YUK LING, Principal Investigator, North District Hospital
Other Study IDs: 2022.354
Record Dates: First submitted 2024-04-09; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Airway Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- coughing with suction: Suction performed on manikin in simulated setting
- coughing with suction covered by surgical mask: Suction performed on manikin in simulated setting
  Interventions: Device: Enclosure barrier
- coughing with suction covered by enclosure tent: Suction performed on manikin in simulated setting
  Interventions: Device: Enclosure barrier

INTERVENTIONS:
Device: Enclosure barrier — Surgical mask & Enclosure tent compared with open suction
  Groups: coughing with suction covered by enclosure tent; coughing with suction covered by surgical mask

SUMMARY:
The aim of the study is to examine the air dispersion pattern and the environmental influence of open airway suction in general ward setting. Secondly, the study is aimed at identifying a simple & practical enclosure device in general ward. Suction will be performed in manikin in supine lying.

Nasopharyngeal suction will be performed by physiotherapist with working experience more than 1 years. Besides, surgical mask & enclosure tent will be adopted as the enclosure barrier device in this study.

Research Question

1. To assess the extent of the environmental contamination during coughing and simulated airway suction
2. To measure the air particle count during coughing and simulated open airway suction.
3. To evaluate how effective the enclosure barrier in reducing the air particle dispersion during open airway suction.

ELIGIBILITY:
Inclusion Criteria:

* physiotherapists with working experience more than one year

Exclusion Criteria:

* physiotherapists with working experience less than one year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Registered physiotherapist
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Air particle count | one minute
  The calibrated sizes are 0.3, 0.5. 1.0, 2.0, 5.0 and 10 microns

SECONDARY OUTCOMES:
A fluorescent Dye | one minute
  The extent and area of the fluorescent dye spreading are measured

CONTACTS AND LOCATIONS:
Overall Officials: Connie TO, Msc, Principal Investigator — NDH
Locations (1):
- North District Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No